CLINICAL TRIAL: NCT06551948
Title: RandomisEd PlAcebo ControlLed TrIal of MethylceILulose or PSyllium on FermentaTion of Inulin Assessed Using a Gas Sensing Capsule (REALISTIC)
Brief Title: Effect of MethylceIlulose or Psyllium on Fermentation of Inulin Assessed Using a Gas Sensing Capsule
Acronym: REALISTIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: University of East Anglia (Other)
Responsible Party: Principal Investigator, Robin Spiller, Professor of Gastroenterology, University of Nottingham
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: FMHS 64-1123
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2024-08

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Psyllium; Methylcellulose; maltodextrin; Inulin

STUDY DESIGN:
Intervention Model Description: 3 way cross over
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Test meals in opaque plastic bags
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Psyllium (Experimental): 15 g psyllium
  Interventions: Dietary Supplement: psyllium; Dietary Supplement: inulin
- methylcellulose (Experimental): 15 g methylcellulose
  Interventions: Dietary Supplement: methylcellulose; Dietary Supplement: inulin
- Maltodextrin (Placebo Comparator): 15 g maltodextrin
  Interventions: Dietary Supplement: maltodextrin; Dietary Supplement: inulin

INTERVENTIONS:
Dietary Supplement: psyllium — 15 g psyllium
  Arms: Psyllium
Dietary Supplement: methylcellulose — 15 gm methylcellulose
  Arms: methylcellulose
Dietary Supplement: maltodextrin — 15 g maltodextrin
  Arms: Maltodextrin
Dietary Supplement: inulin — 15g inulin

SUMMARY:
The investigators plan to measure the local (in vivo) production of hydrogen when methylcellulose is ingested, to see if the investigators can show a shift of the site of fermentation to the distal colon.

The investigators will achieve this using the Atmo pill, a recently developed ingestible gas-sensing wireless capsule manufactured by Atmo Biosciences. The pill is very similar in appearance and dimensions (26·8 mm long by 11·7 mm in diameter) to the Smart Pill, an FDA approved wireless capsule which measures local pH, which has been widely and safely used for over a decade. The Smart Pill is recommended for transit measurement by the American ACG Clinical Guidelines on Gastroparesis 3. The Atmo pill differs from the Smart Pill in measuring hydrogen and carbon dioxide within the colonic lumen rather than pH. The pill emits a radio signal to a small device worn by the participant to record the measurements periodically 4.

DETAILED DESCRIPTION:
Aim

This pilot study aims to test the hypothesis that a gel of either methylcellulose or psyllium incorporating inulin will delay colonic fermentation compared to inulin combined with placebo (maltodextrin), resulting in an increase in colonic hydrogen concentration in the distal colon as measured by the Atmo pill.

Objective

The primary objective of this pilot is to quantify in vivo the hydrogen gas produced from colonic fermentation post ingestion. Previous studies have measured hydrogen concentration from breath analysis to infer colonic fermentation progression, however the Atmo pill will allow for direct measurement throughout colonic transit. By dividing the mean colonic hydrogen gas production into time quartiles, the investigators can better associate which region of the colon the fermentation is taking place (i.e., 4th quartile to represent distal colon region).

Secondary Objectives

Mean colonic hydrogen% in each quarter of colonic transit.

Mean colonic carbon dioxide% in each quarter of colonic transit.

Colon transit time (CTT) determined from Atmo pill.

Small bowel transit time (SBTT) of Atmo pill to caecum.

Area under curve (AUC) of breath hydrogen and methane for period 0 - 24hr.

Orocecal transit time (OCTT) from breath analysis.

Whole gut transit time assessed by blue muffin test.

Gas production over 48 hours incubation in vitro model of colon using participants stool samples (in collaboration with Quadram Institute).

Metabolite production (short chain fatty acids) using same in vitro model of colon (in collaboration with Quadram Institute).

Analysis of microbiota in participants stool using 16sRNA gene (in collaboration with Quadram Institute).

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent.
* Scoring ≤5 (i.e., mild, or less) for symptoms of flatulence, bloating, abdominal pain, loose stool, and hard stool in previous 2 weeks using a modified Gastrointestinal Symptom Rating Scale (5).
* Agrees to consume the meals provided.
* Agrees to not smoke during the breath hydrogen sampling period.

Exclusion Criteria:

* Pregnancy, lactating, or planning pregnancy during the course of the investigation declared by candidate.
* History declared by the candidate of pre-existing gastrointestinal disorder that may affect bowel function.
* Contraindications to Atmo capsule including swallowing disorders, suspected or known strictures or GI surgery within last 3 months or consuming Proton Pump Inhibitors (full details see Atmo manual)
* For any reason, unable to wear or maintain close proximity to (no greater than 1.5 m) the personal receiver which logs the data measured from the Atmo pill for the duration of its whole gut transit.
* Reported history of previous resection of the oesophagus, stomach, or intestine (excluding appendix).
* Intestinal stoma.
* Any medical condition making participation potentially compromising participation in the study e.g., diabetes mellitus, respiratory disease limiting ability to use breath hydrogen analyser, known intolerance to one of the test substances.
* Has a body mass index (BMI) value less than 18.5 or greater than 35.
* Will not agree to follow dietary and lifestyle restrictions required.
* Unable to stop drugs known to alter GI motility including mebeverine, opiates, monoamine oxidase inhibitors, phenothiazines, benzodiazepines, calcium channel antagonists for the duration of the study (Selective serotonin reuptake inhibitors, low dose tricyclic antidepressants, antihistamines, and oral contraceptive pill will be recorded in the CRF but will not be an exclusion criteria).
* Participants who are taking antibiotics or probiotics as it might alters gut microbiota.
* Poor understanding of English language.
* Participation in night shift work the week prior to the study day. Night work is defined as working between midnight and 6.00 AM.
* Anyone who in the opinion of the investigator is unlikely to be able to comply with the protocol e.g., cognitive dysfunction, chaotic lifestyle related to substance abuse.
* Having taken part in a research study in the last 3 months involving invasive procedures or an inconvenience allowance. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Colonic hydrogen per quarter of colonic transit | up to 4 days
  mean hydrogen as % of colonic gas during the 4 quarters of colonic transit

SECONDARY OUTCOMES:
carbon dioxide gas production | up to 4 days
  carbon dioxide as % of colonic gas from colonic fermentation post-ingestion of fibre gel drink ll over each quartile of colonic transit (AUC Q1, Q2, Q3, Q4)

OTHER OUTCOMES:
Breath hydrogen | 0-6 hours
  Area under curve (AUC) from time 0-6 hours of breath hydrogen (ppm.hours)
Regional transit times (hours) of Atmo pill; | up to 4 days

CONTACTS AND LOCATIONS:
Locations (1):
- Nottingham Digestive Disease Centre, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No